CLINICAL TRIAL: NCT04048304
Title: Short Post-surgical Antibiotic Therapy in Spine Infections - a Pro-spective, Randomized, Unblinded, Non-inferiority Trial
Brief Title: Short Post-surgical Antibiotic Therapy in Spine Infections - a Prospective, Randomized, Unblinded, Non-inferiority Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SASI
Record Dates: First submitted 2019-07-12; First posted 2019-08-07 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Amoxicillin-Potassium Clavulanate Combination; Vancomycin

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short antibiotic therapy (Experimental): 3 weeks of antibiotic therapy with no implant left in place 6 weeks of antibiotic therapy with implant left in place
  Interventions: Drug: duration of standard antibiotic therapy
- long antibiotic therapy (Active Comparator): 6 weeks of antibiotic therapy with no implant in place 12 weeks of antibiotic therapy with implant left in place
  Interventions: Drug: duration of standard antibiotic therapy

INTERVENTIONS:
Drug: duration of standard antibiotic therapy — antibiotic therapy for spine infections. 3 vs 6 weeks if no implant left in place. 6 vs 12 weeks if implant left in place. The antibiotic agents used are officially indicated for orthopedic infections, including spine infections and available in Switzerland since decades. Standard dosing will be applied and only modified according to the patient's co-morbidities, intolerances and weight.
  Other Names: Co-amoxiclav, vancomycin

SUMMARY:
We implement a prospective, randomized, unblinded, non-inferiority trial regarding the duration of systemic, targeted antibiotic therapy after the first surgical debridement for spine infection; randomizing 1:1 between

1. Six and twelve weeks of antibiotic therapy if there is an implant left in place
2. Three and six weeks of antibiotic therapy if there is no implant left

ELIGIBILITY:
Inclusion Criteria:

* Spine surgery and intraoperative debridement with any technique
* At least 12 months of scheduled follow-up from hospitalization
* Bacterial spine infection of any nature, independently of implants or co-morbidities

Exclusion Criteria:

* Mycobacterial, fungal, nocardial, and Actinomyces infections in the spine
* Non-resected cancer in the infection site
* Bone marrow or recent solid organ transplant patient (Recent: <5 years)
* Any other infection in the patient requiring more than 6 weeks of antibiotic therapy
* More than three intraoperative debridements performed for spine infection
* Absence of at least one surgical intraoperative debridement of infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission of infection at 12 months after treatment | 12 months after treatment
  no clinical and microbiological recurrences

SECONDARY OUTCOMES:
costs | up to 12 months
  total costs for treatment of infection
duration of sick leave | up to 12 months
  duration of sick leave for treatment of infection
length of hospital stay | up to 12 months
  number of days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uckay, PD Dr med, Study Director — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
identifying IPD will not be shared with other Researchers

REFERENCES:
- [Derived] Zendeli F, Jedrusik A, Schaefer RO, Albrecht D, Betz M, Waibel FWA, Grober T, Kuhne N, Konneker S, Uckay I. Pathogen-Specific Risk for Iterative Surgical Debridement in Orthopedic Infections: A Prospective Multicohort Analysis. J Clin Med. 2025 Dec 10;14(24):8750. doi: 10.3390/jcm14248750. PMID 41464652
- [Derived] Betz M, Uckay I, Schupbach R, Grober T, Botter SM, Burkhard J, Holy D, Achermann Y, Farshad M. Short postsurgical antibiotic therapy for spinal infections: protocol of prospective, randomized, unblinded, noninferiority trials (SASI trials). Trials. 2020 Feb 6;21(1):144. doi: 10.1186/s13063-020-4047-3. PMID 32028985

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04048304/SAP_000.pdf